CLINICAL TRIAL: NCT02673060
Title: A Phase 1 Multicenter, Open-label, Dose-escalation Trial of MBC-11, an Etidronate-ara-C Conjugate in Patients With Malignant Tumors With Cancer-induced Bone Disease (CIBD)
Brief Title: A Trial of MBC-11 in Patients With CIBD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Osteros Biomedica Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OB-MBC-01
Record Dates: First submitted 2016-01-22; First posted 2016-02-03 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Bone Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dose escalation of MBC-11 (Experimental): MBC-11 was administered in 5 consecutively recruited cohort in dose 0.5 mg/kg, 1 mg/kg, 2.5 mg/kg, 5 mg/kg,10 mg/kg accordingly. The dose escalation is aimed at determining the maximum tolerated dose (MTD)
  Interventions: Drug: MBC-11

INTERVENTIONS:
Drug: MBC-11 — 0.5 mg/kg-10 mg/kg , IV (in the vein) on day 1-5 of each 28 day cycle. Number of cycles: 2, in case of partial metabolic reaction or stable metabolic reaction - up to 4.

SUMMARY:
This study evaluates MBC-11 (a conjugate of a bone-targeting vehicle (etidronate) and a cytostatic agent [ara-C] in patients with malignant tumors with CIBD. This is a first use in human.

DETAILED DESCRIPTION:
A standard "3+3" dose escalation design to determine Maximum Tolerated Dose with consecutive different dose level cohort recruitment.

The following dose levels to be investigated: 0.5 mg/kg, 1.0 mg/kg, 2.5 mg/kg, 5.0 mg/kg, 10 mg/kgm 20 mg/kg. The study for each patient consists of 14-days screening period, single dose administration of MBC-11 followed by 7-day safety monitoring and then 2 cycles of multiple use of MBC-11 (28 days each cycle, study drug is administered at Days1-5). In case of partial metabolic reaction/stable metabolic reaction therapy maybe prolonged up to 4 cycles (at investigator and sponsor consideration)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant tumor (breast cancer, prostate cancer etc)
* Bone metastases, documented by radiographs, bone scan
* No available standard chemotherapy or no indication for chemotherapy at the time of screening
* Eastern Cooperative Oncology Group [ECOG] status 0-2
* Adequate bone marrow function (hemoglobin ≥ 9 g/dL with or without transfusion requirement, absolute neutrophil count ≥ 1500/mm3, and platelets ≥ 75,000/mm3)
* Adequate liver function (bilirubin ≤ 2 x Upper Limit of Normal [ULN], Alanine aminotransferase [ALT] ≤ 2.5 x ULN).
* Adequate renal function (creatinine ≤ 1.5 x ULN) and creatinine clearance ≥ 50 mL/min [measured or calculated by nomogram]).

Exclusion Criteria:

* Systemic chemotherapy and/or investigational therapy within the previous 4 weeks
* Fracture ≤ 6 month prior the inclusion in the study
* Brain metastasis
* Serum calcium levels < 8.5 mg/dL (< 2.2 mmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | up to 20 weeks
  evaluation of adverse events, physical examination, laboratory parameters
Dose Limiting Toxicity [DLT] | up to 20 weeks
  dose limiting toxicity is graded according to NCI CN CFT version 4
Maximum tolerated dose | up to 20 weeks

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] of MBC-11 | 5 weeks
  Cmax will be evaluated during Cycle 1
Pharmacodynamic parameters | up to 20 weeks
  Levels of bone turnover markers is measured
Fluorodeoxyglucose positron emission tomography-computed tomography [FDG PET-CT] response after cycle 2 and cycle 4 therapy | up to 20 weeks
  Response rate according to Positrone Emission Tomography Response Criteria in Solid Tumors [PERCIST] criteria using FDG PET/CT
Maximum Plasma Concentration [Cmax] of etidronate | 5 weeks
  pharmacokinetics [PK] assessment of MBC-11 metabolite
Maximum Plasma Concentration [Cmax] of ara-U | 5 weeks
  PK assessment of MBC-11 metabolite
Peak time [Tmax] for MBC-11 | 5 weeks
  PK parameters assessment of study drug
Peak time [Tmax] for etidronate | 5 weeks
  PK assessment of MBC-11metabolite

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zinnen SP, Karpeisky A, Von Hoff DD, Plekhova L, Alexandrov A. First-in-Human Phase I Study of MBC-11, a Novel Bone-Targeted Cytarabine-Etidronate Conjugate in Patients with Cancer-Induced Bone Disease. Oncologist. 2019 Mar;24(3):303-e102. doi: 10.1634/theoncologist.2018-0707. Epub 2018 Nov 9. PMID 30413669